CLINICAL TRIAL: NCT02143089
Title: Evaluation OF Use Versus Non Use of Urinary Catheterization During Second Elective Caesarean Delivery
Brief Title: Catheterization During Second Elective Caesarean Delivery
Acronym: CDSECD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Salwa Said Ali Wahba, Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HSM28-10-12
Record Dates: First submitted 2014-05-06; First posted 2014-05-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Wound Infection
Keywords: CCSWI
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Use of urinary catheterization in Cesarean section
  Interventions: Device: Foley's Catheter
- Group 2 (No Intervention): NO urinary catheterization during Cesarean section

INTERVENTIONS:
Device: Foley's Catheter — Urinary tract infection inpatient catheterized versus non catheterized
  Arms: Group 1

SUMMARY:
Use versus non use of urinary catheterization during Second Elective caesarean delivery:

DETAILED DESCRIPTION:
Evaluation OF use versus non use of urinary catheterization during Second Elective caesarean delivery:by urine analysis 24 hours postoperative to exclude urinary tract infection.

ELIGIBILITY:
inclusion criteria

* pregnant females who will undergo second elective caesarean section at full term pregnancy (38:41 weeks gestational age).

Exclusion Criteria:

* Women with history of more than one previous caesarean Section.
* Women with history of a tonic postpartum hemorrhage.
* Women with Urinary tract infection in present pregnancy.
* Women with diabetes mellitus in present pregnancy.
* Women with medical disorder in present pregnancy that obligate monitoring of urine output during and after caesarean section, such as severe pre-eclampsia or renal disease with pregnancy.
* Emergency caesarean section

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-08 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Urine analysis to diagnosed urinary tract infection by leucocytes more than 10 per high power field | participants will be followed for the duration of urinary tract infection,an expected average 2 days.

CONTACTS AND LOCATIONS:
Overall Officials: Amr Helmy, Master, Principal Investigator — Ain Shams University
Locations (1):
- AinShamsU, Cairo, Egypt